CLINICAL TRIAL: NCT00424827
Title: A Phase II Trial of Cetuximab, Gemcitabine, 5-Fluorouracil and Radiation Therapy in Locally Advanced Non-metastatic Pancreatic Adenocarcinoma
Brief Title: A Trial of Chemo & Radiation Therapy for Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UM200602
Record Dates: First submitted 2007-01-18; First posted 2007-01-22 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer, gemcitabine, 5-FU, cetuximab, radiation
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Fluorouracil; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine/Fluorouracil with External Beam Radiation (Experimental): This protocol will assess the antitumor activity of Gemcitabine/Fluorouracil with External Beam Radiation in patients with non-metastatic, locally advanced pancreatic carcinoma.
  Interventions: Drug: Gemcitabine/Fluorouracil with External Beam Radiation

INTERVENTIONS:
Drug: Gemcitabine/Fluorouracil with External Beam Radiation — This protocol will assess the antitumor activity of gemcitabine (200 mg/m2 per week) and cetuximab (400mg/m2 loading dose followed by 250 mg/m2 weekly) when given with continuous infusion 5-FU (200 mg/m2/day/M-F) and daily concurrent external beam radiation therapy (50.4 Gy) in patients with non-metastatic, locally advanced pancreatic carcinoma.
  Other Names: EGFR Expression; Cetuximab & Radiosensitization of Cetuximab

SUMMARY:
This is an open-label, non-randomized, combination study of cetuximab, gemcitabine, 5-FU, and external beam radiotherapy in patients with locally advanced, non-metastatic pancreatic cancer.

DETAILED DESCRIPTION:
During cycle I (chemoradiation), gemcitabine (200 mg/m2) and cetuximab 400mg/m2 initial dose followed by 250mg/m2 IV weekly will be given with continuous infusion 5-FU (200 mg/m2/day) delivered 5 of every 7 days and concurrent external beam radiation therapy. Cetuximab, gemcitabine and 5-FU will begin on the first week of external beam radiotherapy and will continue throughout the course of external beam radiation therapy, and will be discontinued following the conclusion of external beam radiation therapy. All patients will have a central venous access device placed to facilitate chemotherapy administration.

During cycles 2 through 5 (chemotherapy), gemcitabine will be administered at a dose of 1000 mg/m2 over 30 minutes followed by cetuximab at a dose of 250mg/m2 over 30 minutes weekly for 3 weeks followed by one-week rest for four cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of pancreatic adenocarcinoma is required.
* Only patients with unresectable, non-metastatic tumors are eligible.
* Documentation of disease extent by endoscopic ultrasound and either laparotomy or laparoscopy must be performed within 42 days of registration.
* All patients will also be assessed by chest x-ray and abdominal-pelvic CT scan.
* Confirmation of palliative surgical bypass at the time of laparotomy or whether a biliary stent was placed will be requested.
* Disease must be locoregional and not amenable to surgery based on one or more of the following criteria:

  * size of pancreatic tumor > 5 cm.
  * lymph nodes (bulky, > 2 cm, but within a radiation port)
  * vascular involvement or impingement of major vessels (superior mesenteric artery, superior mesenteric vein, portal vein, hepatic artery).
  * invasion into the adjacent structures.
* Patients with either measurable or evaluable disease are eligible.
* Patients with evidence of peritoneal seeding by malignancy are not eligible for the study.
* Patients with other evidence of metastatic disease are not eligible.
* Patients with concurrent malignancy of any site, except limited basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, are ineligible.
* Patients with any other malignancy within 5 years of study entry, except curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, are ineligible.
* Patients may not have had prior therapy for carcinoma of the pancreas, nor prior abdominal radiation therapy.
* Age > 18 years.
* CTC performance status < 2.
* No myocardial infarction in the past six months.
* No major surgery in the past two weeks.
* No uncontrolled serious medical or psychiatric illness.
* Required Initial Laboratory Data:

  * Total bilirubin < 2.0 mg/dl
  * AST < 3x upper limits of normal.
  * Serum creatinine < 2.0 mg/dl
  * WBC > 3,000/mm3 (ANC>1500/mm3)
  * Platelets > 100,000 mm3
  * CA 19-9
* Required Diagnostic procedures:

  * Chest X-ray
  * Abdominal pelvic CT scan
  * EUS
  * Staging laparoscopy or staging laparotomy

Exclusion Criteria:

Enrollment in this trial will be limited to patients for whom protocol therapy is safe and appropriate. Physicians should consider the risks and benefits of therapy together with all relevant medical and other considerations in deciding whether this protocol is appropriate for a particular patient. Specific considerations include:

* Psychiatric illness which would prevent the patient from giving informed consent.
* Serious medical illness such as uncontrolled infection, severe cardiovascular disease including recent (< 6 months) myocardial infarction or uncontrolled congestive heart failure, or other serious illness which would limit anticipated survival to < 12 weeks.
* Protocol treatment would pose significant risk to an unborn child. Pregnant women should not be enrolled, and women of child-bearing age should be strongly encouraged to practice effective birth control during and for three months after the trial.
* Inability to swallow medication. Patients should have adequate, unassisted oral intake.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Venu Bathini, MD, Principal Investigator — University of Massachusetts, Worcester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 2006 and 2011, twenty-six patients were screened and eleven of them were enrolled in the study. Most common reasons for screen failures were having resectable disease, metastatic disease or co-morbidity. Ten patients were able to tolerate and complete cycle 1 of chemoradiotherapy.
Pre-assignment Details: Most common reasons for screen failures were having resectable disease, metastatic disease or co-morbidity. A minority of patients present with localized disease. Surgical resection only hope for long-term survival. Locally advanced pancreatic cancer is defined as surgically unresectable, but has no evidence of distant metastases.
Groups:
- Single Arm: This protocol will assess the antitumor activity of gemcitabine (200 mg/m2 per week) and cetuximab (400mg/m2 loading dose followed by 250 mg/m2 weekly) when given with continuous infusion 5-FU (200 mg/m2/day/M-F) and daily concurrent external beam radiation therapy (50.4 Gy) in patients with non-metastatic, locally advanced pancreatic carcinoma.
  Gemcitabine/Fluorouracil with External Beam Radiation: This protocol will assess the antitumor activity of gemcitabine (200 mg/m2 per week) and cetuximab (400mg/m2 loading dose followed by 250 mg/m2 weekly) when given with continuous infusion 5-FU (200 mg/m2/day/M-F) and daily concurrent external beam radiation therapy (50.4 Gy) in patients with non-metastatic, locally advanced pancreatic carcinoma.
Period: Overall Study
Arm/Group | Single Arm
Started | 11
Completed | 10
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Subjects with non-metastatic, locally advanced pancreatic adenocarcinoma. Following neoadjuvant treatment, subjects were re-evaluated for response and surgical candidacy with restaging scans.
Groups:
- This Was a Prospective, Single Arm, Open Label Pilot Phase II: "A Phase II Trial of Cetuximab, Gemcitabine, 5-Fluorouracil, and Radiation Therapy in Locally Advanced Nonmetastatic Pancreatic Adenocarcinoma"
  This protocol will assess the antitumor activity of gemcitabine (200 mg/m2 per week) and cetuximab (400mg/m2 loading dose followed by 250 mg/m2 weekly) when given with continuous infusion 5-FU (200 mg/m2/day/M-F) and daily concurrent external beam radiation therapy (50.4 Gy) in patients with non-metastatic, locally advanced pancreatic carcinoma.
  Locally advanced pancreatic cancer is defined as surgically unresectable, but has no evidence of distant metastases. The purpose of this study is to evaluate the efficacy and safety of cetuximab in combination with gemcitabine and 5-FU along with radiation therapy in locally advanced non-resectable, pancreatic adenocarcinoma, using progression free survival as the primary end point.
Arm/Group | This Was a Prospective, Single Arm, Open Label Pilot Phase II
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 66 [48 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival of Patients With Locally Advanced Pancreatic Cancer Treated With Concurrent Gemcitabine, 5-FU, Cetuximab and External Beam Radiation Therapy.
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 1-year
Population: Must have histologic confirmation of pancreatic adenocarcinoma with measurable disease per RECIST criteria, with locoregional disease not amenable to surgery were enrolled: based on(1) size of the tumor, 5cm; (2) lymph nodes; (3) vascular involvement or impingement on major vessels; and (4) invasion into the adjacent structures.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Gemcitabine/Fluorouracil With External Beam Radiation:: Progression-free survival
Arm/Group | Gemcitabine/Fluorouracil With External Beam Radiation:
Number analyzed (Participants) | 11
months | 7.17 [2.53 to 18.43]

2. Secondary Outcome: Biomarker Response to Chemoradiation Therapy
Description: 20% decrease in biomarker (CA19-9) from baseline
Time Frame: 1-year
Population: Biomarker response (CA19-9) as defined by at least a 20% decrease from baseline
Measure: Number; unit: participants
Arm/Group | Gemcitabine/Fluorouracil With External Beam Radiation:
Number analyzed (Participants) | 10
participants | 7

3. Secondary Outcome: Resection Rate
Time Frame: 1-Year
Population: 4 subjects underwent resection after treatment
Measure: Number; unit: participants
Arm/Group | Gemcitabine/Fluorouracil With External Beam Radiation:
Number analyzed (Participants) | 11
participants | 4

4. Secondary Outcome: Overall Survival
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine/Fluorouracil With External Beam Radiation:
Number analyzed (Participants) | 11
months | 17 [7.1 to 27.6]

5. Secondary Outcome: Toxicity Associated With This Regimen.
Time Frame: 1-Year
Measure: Number; unit: participants
Arm/Group | Gemcitabine/Fluorouracil With External Beam Radiation:
Number analyzed (Participants) | 11
participants | 2

ADVERSE EVENTS:
Time Frame: 3 years
Description: Subjects were evaluated every 3 months for 1 year, then every 6 months for an additional 2 years
Groups:
- Gemcitabine/Fluorouracil With External Beam Radiation: antitumor activity of gemcitabine (200 mg/m2 per week) and cetuximab (400mg/m2 loading dose followed by 250 mg/m2 weekly) when given with continuous infusion 5-FU (200 mg/m2/day/M-F) and daily concurrent external beam radiation therapy (50.4 Gy) in patients with non-metastatic, locally advanced pancreatic carcinoma.
Arm/Group | Gemcitabine/Fluorouracil With External Beam Radiation
Serious Adverse Events (participants affected / at risk) | 4/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine/Fluorouracil With External Beam Radiation (N=11)
Cardiac Dysrhythmia (Cardiac disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) — Subject was hospitalized with severe nausea
radiation-related duodenitis, biliary obstruction (Gastrointestinal disorders) | 1 (1)
Dehydration, biliary obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine/Fluorouracil With External Beam Radiation (N=11)
Lymphopenia (Blood and lymphatic system disorders) | 10 (17)
Diarrhea (Gastrointestinal disorders) | 8 (17)
Hypoalbuminemia (Blood and lymphatic system disorders) | 8 (10)
hypocalcemia (Blood and lymphatic system disorders) | 8 (10)
nausea (Gastrointestinal disorders) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No